CLINICAL TRIAL: NCT02685150
Title: The Role of Endoscopic Tri-Modal Imaging in Distinguishing Functional Dyspepsia From Reflux Disease
Brief Title: Endoscopic Tri-Modal Imaging to Distinguish Functional Dyspepsia From Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Weifeng Wang, MD, Associate Professor, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S2015-086-02
Record Dates: First submitted 2016-01-19; First posted 2016-02-18 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Gastroesophageal Reflux Disease; Dyspepsia; Bile Reflux
Keywords: Endoscopic Tri-Modal Imaging; Gastric juice; Functional dyspepsia; Acid reflux disease; Bile reflux
MeSH Terms: conditions — Gastroesophageal Reflux; Dyspepsia; Bile Reflux | interventions — Omeprazole; Proton Pump Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Functional dyspepsia (Experimental): Participants are to undergo Endoscopic Tri-Modal Imaging, Omeprazole test and Analysis of gastric juice and those who fulfill with Rome III criteria for functional dyspepsia are to be classified into this group.
  Interventions: Device: Endoscopic Tri-Modal Imaging; Drug: Omeprazole; Other: Analysis of gastric juice
- Acid reflux disease (Experimental): Participants are to undergo Endoscopic Tri-Modal Imaging, Omeprazole test and Analysis of gastric juice. Participants with acid reflux are to confirmed by Omeprazole test, one kind of proton-pump inhibitor (PPI) tests.
  Interventions: Device: Endoscopic Tri-Modal Imaging; Drug: Omeprazole; Other: Analysis of gastric juice
- Bile reflux disease (Experimental): Participants are to undergo Endoscopic Tri-Modal Imaging and Analysis of gastric juice. Participants with bile reflux are to be confirmed by Analysis of gastric juice.
  Interventions: Device: Endoscopic Tri-Modal Imaging; Other: Analysis of gastric juice
- Health volunteers (Experimental): Health volunteers for routine checkup. Participants are to undergo Endoscopic Tri-Modal Imaging as well as Analysis of gastric juice and those who show no abnormal findings are to be classified into this group.
  Interventions: Device: Endoscopic Tri-Modal Imaging; Other: Analysis of gastric juice

INTERVENTIONS:
Device: Endoscopic Tri-Modal Imaging — Endoscope that combines white light imaging (WLI) with autofluorescence imaging (AFI) and narrow band imaging (NBI).
Drug: Omeprazole — Omeprazole is one kind of proton-pump inhibitors. All participants undergo standard proton-pump inhibitor (PPI) tests for two weeks with Omeprazole, 20mg twice a day.
  Other Names: proton-pump inhibitor (PPI)
  Arms: Acid reflux disease; Functional dyspepsia
Other: Analysis of gastric juice — Analysis of gastric juice including routine, biochemical and microbiological analysis.
  Other Names: Routine,biochemical, microbiological analysis

SUMMARY:
Endoscopic Tri-Modal Imaging which combines Narrow-band Imaging(NBI), Autofluorescence Imaging (AFI) and White-light Imaging (WLI) could be used to identify the indistinct changes in the gut caused by reflux disease,either acid reflux or bile reflux, which make it possible to differentiate reflux disease from functional dyspepsia (FD).

DETAILED DESCRIPTION:
Functional dyspepsia (FD) and acid/bile reflux disease are common. These diseases share similar clinical manifestations. Individuals with functional dyspepsia (FD) often present upper abdominal pain or discomfort, bloating, early satiety, loss of appetite, and no organic factors underlie it. Individuals suffering from acid/bile reflux disease often complain heartburn, upper abdominal burning or discomfort. What is more, there are always no specific changes on traditional endoscopy that can be used to differentiate these diseases (except erosive esophagitis). Though proton-pump inhibitor (PPI) test is frequently applied to confirm the diagnosis of acid reflux disease, but certain amounts of individuals with gastroesophageal reflux disease (GERD) do not show favorable response to PPI test. In order to make a distinction of these diseases, esophageal pH-metry is needed, however it is not always available in most clinics. Recent data showed that new endoscopic technology such as Endoscopic Tri-Modal Imaging could demonstrate indistinct lesions caused by GERD which are not detectable by standard endoscopy, subsequently improve endoscopic diagnosis of these diseases. In addition, simultaneous analysis of gastric juice can help to determine whether bile reflux is present or not. As it is known, pathologic refluxes underlie not functional dyspepsia but acid/bile reflux disease. Hence, it is hypothesized that Endoscopic Tri-Modal Imaging in combination with simultaneous analysis of gastric juice could be used to differentiate functional dyspepsia from acid/bile reflux disease.

ELIGIBILITY:
Inclusion Criteria:

* symptoms suggestive of GERD or dyspepsia.
* Presence of symptom for longer than 6 month
* Provision of written informed consent

Exclusion Criteria:

* Any known upper GI disease, other than reflux esophagitis
* Active or healing gastroduodenal ulcer (except scars)
* History of esophageal or gastric surgery.
* Clinically significant heart, lung, liver or kidney disease
* Allergy to proton-pump inhibitor
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2016-01; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Numbers of participants with abnormal endoscopic findings and positive Omeprazole tests | one month
  Numbers of participants with abnormal endoscopic findings are used to calculate the diagnostic Value of Endoscopic Tri-Modal Imaging in Distinguishing Functional Dyspepsia and Reflux Disease, including specificity, sensitivity and accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Guoquan Ren, Ph.D., Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Data are available from the W Wang, MD.

REFERENCES:
- [Background] Talley NJ. Functional (non-ulcer) dyspepsia and gastroesophageal reflux disease: one not two diseases? Am J Gastroenterol. 2013 May;108(5):775-7. doi: 10.1038/ajg.2013.102. PMID 23644963
- [Result] Wang W, Uedo N, Yang Y, Peng L, Bai D, Lu Z, Fan K, Wang J, Wang X, Zhao Y, Yu Z. Autofluorescence imaging endoscopy for predicting acid reflux in patients with gastroesophageal reflux disease. J Gastroenterol Hepatol. 2014;29(7):1442-8. doi: 10.1111/jgh.12566. No abstract available. PMID 25587615